CLINICAL TRIAL: NCT01711775
Title: A Single-center, Non-randomized, Open-label Study to Assess the Pharmacokinetics of Aleglitazar (RO0728804) After Administration of Single and Multiple Oral Doses of 150 µg Tablet in Healthy Chinese Subjects
Brief Title: A Pharmacokinetic Study of Aleglitazar in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP25230
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar

ARMS (1):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar

INTERVENTIONS:
Drug: aleglitazar — Single oral dose Day 1, repeated oral dose once daily Days 5-14

SUMMARY:
This single-center, non-randomized, open-label study will assess the pharmacokinetics of aleglitazar after administration of single and multiple oral doses in healthy Chinese volunteers. Subjects will receive a single oral dose of aleglitazar on Day 1 and repeated oral doses once daily from Day 5 to Day 14. Anticipated time on study, including screening and a 2-week follow-up, is up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male Chinese volunteers, 18 to 45 years of age inclusive at screening
* Subjects have to be healthy as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory measurements performed at screening
* Body mass index (BMI) 19 to 24 kg/m2 inclusive
* Female subjects who are not surgically sterile must be willing to use effective method of contraception as defined by protocol throughout the study and for 30 days after the last dosing

Exclusion Criteria:

* Any significant allergic reactions or multiple allergies
* Diagnosed or treated malignancy (except for treated cases of basal skin cancer or in situ carcinoma of the cervix) within the past 5 years
* Any major illness within 2 months prior to first dosing or febrile illness within 14 days prior to first dosing
* Positive for hepatitis B, hepatitis C or HIV infection
* Any clinically relevant history of alcohol and/or other substance abuse or addiction within the last 2 years
* Pregnant or lactating women, or women who have a positive pregnancy test
* Regular smoker with consumption of more than 10 cigarettes per day or equivalent amount of tobacco
* Participation in an investigational drug or device study within 3 months prior to the first dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Day 14 (steady-state) maximum concentration (Cmax) | Day 14 pre-dose and up to 24 hours post-dose
Pharmacokinetics: Day 14 (steady-state) area under the concentration-time curve (AUC 0-24) | Day 14 pre-dose and up to 24 hours post-dose

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum concentration (Cmax) | 18 days
Single-dose pharmacokinetics: Time to maximum observed plasma concentration (tmax) | up to 5 days
Single-dose pharmacokinetics: Half-life (t1/2) | up to 5 days
Single-dose pharmacokinetics: Area under the concentration-time curve (AUC) | up to 5 days
Pharmacokinetics: Apparent oral plasma clearance (CL/F) | 18 days
Pharmacokinetics: Apparent volume of distribution (VZ/F) | 18 days
Pharmacokinetics: Accumulation index (Rac) | 18 days
Safety: Incidence of adverse events | approximately 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Beijing, China